CLINICAL TRIAL: NCT03284723
Title: A Phase 1 Dose Escalation Study Evaluating the Safety and Tolerability of PF-06804103 in Patients With Human Epidermal Growth Factor Receptor 2 (HER2) Positive and Negative Solid Tumors
Brief Title: PF-06804103 Dose Escalation in HER2 Positive and Negative (Negative Only in Part 2) Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated based on the stage in drug development and assessment of PF-06804103 relative to the leading external competition. The decision was not due to a safety concern.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C0541001; 2017-002538-22 (EudraCT Number)
Record Dates: First submitted 2017-09-01; First posted 2017-09-15 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Breast Neoplasms
Keywords: HER2; PF-06804103; ADC; breast cancer; neoplasms; solid tumors; human epidermal growth receptor 2
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — PF-06804103

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06804103 (Experimental): Study Treatment
  Interventions: Drug: PF-06804103
- PF-06804103+Combination Regimen (Experimental): Study Treatment
  Interventions: Drug: PF-06804103 + Palbociclib +Letrozole

INTERVENTIONS:
Drug: PF-06804103 — Dose Escalation Part - 1A Dose Expansion Part - 2A
  Arms: PF-06804103
Drug: PF-06804103 + Palbociclib +Letrozole — Dose Escalation - Part 1B Dose Expansion - Part 2B
  Arms: PF-06804103+Combination Regimen

SUMMARY:
The study will evaluate the safety, pharmacokinetics and pharmacodynamics of increasing doses of PF-06804103 in patients with HER2 positive and negative breast and gastric cancer (HER2 positive only and gastric were studied in Part 1A only). The study will expand to look at selected doses in patients with HER2 positive and negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* HER2 positive breast cancer or gastric cancer that is resistant to standard therapy or for which no standard therapy is available (Part 1A only)
* HER2 positive and negative breast cancer (Part 2A)
* HER2 negative breast cancer (Part 1B & Part 2B)
* Performance status of 0 or 1
* Adequate bone marrow, kidney and liver function

Exclusion Criteria:

* Known CNS disease including, but not limited to, metastases
* History of exposure to certain cumulative doses of anthracyclines
* Grade 3 or higher hypersensitivity reaction to prior receipt of any antibody therapy
* Active and clinically significant bacterial, fungal, or viral infection
* Abnormal cardiac function defined by a LVEF <50% by ECHO or MUGA
* Patients with previous history or active interstitial lung disease or pulmonary fibrosis, or a history of other clinically significant lung diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- United States (26):
  - Banner-University Medical Center Tucson, Tucson, Arizona
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - UCLA Health (main campus), Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - Santa Monica - UCLA Medical Center and Orthopaedic Hospital, Santa Monica, California
  - UCLA Dept of Medicine - Hematology/Oncology, Santa Monica, Santa Monica, California
  - UCLA Health, Santa Monica, Santa Monica, California
  - Northside Hospital Inc.- GCS/Athens, Athens, Georgia
  - Atlanta Cancer Care - Atlanta, Atlanta, Georgia
  - Northside Hospital, Inc. - GCS/Northside, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital,Inc.-GCS /Blairsville, Blairsville, Georgia
  - Northside Hospital, Inc. - GCS/Canton, Canton, Georgia
  - Atlanta Cancer Care - Cumming, Cumming, Georgia
  - Northside Hospital, Inc.-GCS/Stemmer, Decatur, Georgia
  - Suburban Hematology-Oncology Associates - Duluth, Duluth, Georgia
  - Atlanta Cancer Care - Lake Spivey, Jonesboro, Georgia
  - Suburban Hematology-Oncology Associates- Lawrenceville, Lawrenceville, Georgia
  - Northside Hospital, Inc. - GCS/Macon, Macon, Georgia
  - Northside Hospital, Inc. GCS/Kennestone, Marietta, Georgia
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
- Italy (5):
  - Istituto Clinico Humanitas U. O. Oculistica, Milan, Lombardy
  - Azienda Socio-Sanitaria Territoriale Monza, Monza, MB
  - Fondazione IRCCS, Istituto Nazionale dei Tumori, Milan, MI
  - Divisione di Cardiologia - Istituto Europeo di Oncologia Divisione di Medicina Nucleare, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
- Russia (2):
  - LLC "Clinica UZI 4D", Pyatigorsk, Stavropol Kray
  - Private Healthcare Institution "Clinical hospital "RZD-Medicine" of Saint-Petersburg, Saint Petersburg
- South Korea (6):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Universitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Meric-Bernstam F, Calvo E, Lee KS, Moreno V, Park YH, Rha SY, Chalasani P, Zhong W, Zhou L, Pirie-Shepherd S, Leung ACF, Curigliano G. Safety and Tolerability of a Novel Anti-HER2 Antibody-Drug Conjugate (PF-06804103) in Patients with HER2-Expressing Solid Tumors: A Phase 1 Dose-Escalation Study. Mol Cancer Ther. 2023 Oct 2;22(10):1191-1203. doi: 10.1158/1535-7163.MCT-23-0101. PMID 37420274
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0541001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A (PF-06804103 monotherapy) included Part 1A (dose escalation part) and Part 2A (dose expansion part). Part B (PF-06804103 plus palbociclib and letrozole combination therapy) included Part 1B (dose escalation part).
Pre-assignment Details: In Part 1A, 47 participants were treated at dose levels of PF-06804103 0.15, 0.5, 1.2, 2.0, 3.0, 4.0 and 5.0 mg/kg. In Part 2A, 46 participants were treated at dose levels of PF-06804103 3.0 and 4.0 mg/kg. In Part 1B, 2 participants received PF-06804103 2.0 mg/kg in combination with standard of care (SOC) doses of palbociclib and letrozole. Participants were unique in each part.
Groups:
- PART 1A PF-06804103 0.15 mg/kg: Participants with HER2-positive BC or HER2-positive GC received PF-06804103 at 0.15 mg/kg on Day 1 of each 21-day cycle as an intravenous (IV) infusion. The maximum duration of treatment for Part 1A was approximately 89.3 weeks. HER2 = Human Epidermal Growth Factor Receptor 2; BC = breast cancer; GC = gastric and gastroesophageal cancer.
- PART 1A PF-06804103 0.5 mg/kg: Participants with HER2-positive BC or HER2-positive GC received PF-06804103 at 0.5 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 1A was approximately 89.3 weeks.
- PART 1A PF-06804103 1.2 mg/kg: Participants with HER2-positive BC or HER2-positive GC received PF-06804103 at 1.2 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 1A was approximately 89.3 weeks.
- PART 1A PF-06804103 2.0 mg/kg: Participants with HER2-positive BC or HER2-positive GC received PF-06804103 at 2.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 1A was approximately 89.3 weeks.
- PART 1A PF-06804103 3.0 mg/kg: Participants with HER2-positive BC or HER2-positive GC received PF-06804103 at 3.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 1A was approximately 89.3 weeks.
- PART 1A PF-06804103 4.0 mg/kg: Participants with HER2-positive BC or HER2-positive GC received PF-06804103 at 4.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 1A was approximately 89.3 weeks.
- PART 1A PF-06804103 5.0 mg/kg: Participants with HER2-positive BC or HER2-positive GC received PF-06804103 at 5.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 1A was approximately 89.3 weeks.
- PART 2A PF-06804103 3.0 mg/kg HER2+ BC: Participants with HER2-positive BC in third line (3L) setting received PF-06804103 at 3.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 2A was approximately 49.4 weeks.
- PART 2A PF-06804103 4.0 mg/kg HER2+ BC: Participants with HER2-positive BC in 3L setting received PF-06804103 at 4.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 2A was approximately 49.4 weeks.
- PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC: Participants with HR-positive HER2 IHC
  1+ or IHC 2+/ISH- BC in second line (2L) setting received PF-06804103 at 3.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 2A was approximately 49.4 weeks. HR = hormone receptor; IHC = immunohistochemistry; ISH = in-situ hybridization.
- PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC: Participants with HR-positive HER2 IHC
  1+ or IHC 2+/ISH- BC in 2L setting received PF-06804103 at 4.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 2A was approximately 49.4 weeks.
- PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC: Postmenopausal participants with HR-positive HER2 IHC 1+ or IHC 2+/ISH- BC received PF-06804103 at 2.0 mg/kg once every 14 days in a 28-day cycle as an IV infusion. The maximum duration of treatment for Part 1B was approximately 53.7 weeks.
Period: Overall Study
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Started | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 12 | 15 | 2
Received Treatment | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 12 | 15 | 2
Completed | 1 | 2 | 1 | 3 | 9 | 10 | 3 | 5 | 6 | 7 | 9 | 0
Not Completed | 1 | 0 | 1 | 1 | 7 | 5 | 3 | 0 | 8 | 5 | 6 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5 | 3 | 1 | 0 | 6 | 0 | 3 | 1
Not completed — Other | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC | Total
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 12 | 15 | 2 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.0 (19.8) | 65.5 (0.71) | 58.0 (11.31) | 67.0 (4.69) | 54.5 (11.06) | 53.1 (11.70) | 55.5 (11.33) | 50.8 (6.57) | 50.0 (8.68) | 58.3 (10.36) | 53.8 (11.67) | 53.0 (9.90) | 54.5 (10.74)
Age, Customized [Number; unit: Participants]
  <18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 | 1 | 0 | 0 | 0 | 3 | 4 | 1 | 1 | 5 | 1 | 5 | 0 | 21
  45-64 | 1 | 0 | 1 | 1 | 10 | 8 | 4 | 4 | 8 | 7 | 7 | 2 | 53
  >=65 | 0 | 2 | 1 | 3 | 3 | 3 | 1 | 0 | 1 | 4 | 3 | 0 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2 | 11 | 10 | 4 | 5 | 14 | 12 | 15 | 2 | 77
  Male | 2 | 1 | 1 | 2 | 5 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 6
  Not Hispanic or Latino | 2 | 1 | 2 | 4 | 14 | 14 | 6 | 5 | 14 | 11 | 13 | 2 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 4 | 5 | 1 | 1 | 9 | 1 | 3 | 2 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  White | 1 | 1 | 2 | 2 | 10 | 10 | 5 | 4 | 4 | 11 | 12 | 0 | 62
  More than one race | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cycle 1 (21 Days) Dose-Limiting Toxicities (DLTs) in Part 1A
Description: A DLT was any of the following adverse events(AEs) in the first cycle of treatment (within 21 days of first dose). (1) Hematologic: Grade 4 neutropenia lasting >7 days; febrile neutropenia; Grade >＝3 neutropenic infection; Grade >＝3 thrombocytopenia with bleeding; thrombocytopenia; (2) Non-hematologic: Grade >=3 toxicities that were considered clinically significant; delayed by more than 2 weeks in receiving the next scheduled cycle due to persisting treatment related toxicities; concurrent AST or ALT >3x ULN and total bilirubin >2x ULN; any Grade 5 event.
Time Frame: First cycle, Day 1 up to Day 21
Population: Participants enrolled in Part 1A who received at least 1 dose of study treatment and who did not have major treatment deviations during first cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6
Participants | 0 | 0 | 0 | 0 | 2 | 2 | 0

2. Primary Outcome: Number of Participants Wth Cycle 1 (28 Days) Dose-Limiting Toxicities (DLTs) in Part 1B
Description: A DLT was any of the following adverse events(AEs) in the first cycle of treatment (within 28 days of first dose). (1) Hematologic: including a delay greater than 1 week in administration of the next scheduled dose of study treatment due to persistent treatment-related toxicities; Grade 4 neutropenia lasting >7 days; febrile neutropenia; Grade >=3 neutropenic infection; Grade >=3 thrombocytopenia with bleeding; thrombocytopenia. (2) Non-hematologic: including Grade >=3 toxicities that are considered clinically significant; Grade 3 QTc prolongation despite correction of reversible causes; delayed by >2 week in receiving the next scheduled dose of any study treatment due to persisting treatment-related toxicities; inability to administer at least 80% of the planned palbociclib or letrozole or 100% of the planned PF-06804103 doses during Cycle 1 due to toxicity related to the study treatment; concurrent AST or ALT >3x ULN and total bilirubin >2x ULN; any Grade 5 event.
Time Frame: First Cycle, Day 1 up to Day 28
Population: Participants enrolled in Part 1B who received at least 1 dose of study treatment and who did not have major treatment deviations during first cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 1
Participants | 0

3. Primary Outcome: Number of Participants With All-Causality Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event (SAEs), Treatment-Related TEAEs and SAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs (TEAEs) were defined as those with initial onset or increasing in severity after the first dose of study medication. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. Relatedness to study drug was assessed by the investigator.
Time Frame: From the first dose of study treatment up to a minimum of 28 calendar days after the last dose of study treatment (maximum duration between first and last dose: 89.3 weeks for Part 1A, 49.4 weeks for Part 2A, 53.7 weeks for Part 1B)
Population: All enrolled participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 12 | 15 | 2
Participants
  Number of Participants with all-causality TEAEs | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 12 | 15 | 2
  Number of Participants with all-causality SAEs | 1 | 0 | 0 | 1 | 7 | 5 | 4 | 2 | 6 | 5 | 7 | 0
  Number of Participants with treatment-related TEAEs | 1 | 1 | 1 | 4 | 15 | 15 | 6 | 5 | 14 | 10 | 15 | 2
  Number of Participants with treatment-related SAEs | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 5 | 1 | 5 | 0

4. Primary Outcome: Number of Participants With Laboratory Abnormalities-Hematology
Description: Participants who experienced hematology laboratory test abnormalities were summarized according to worst toxicity grade observed for each hematology laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03 (Grade 0: no change from normal or reference range; Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated). This outcome measure calculated the number of participants with hematology laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above, including the following parameters: anemia, INR increased, lymphocyte count decreased, neutrophil count decreased, white blood cell decreased.
Time Frame: From baseline to end of treatment (maximum treatment duration: 89.3 weeks for Part 1A, 49.4 weeks for Part 2A, 53.7 weeks for Part 1B)
Population: Participants who had at least one on-treatment assessment for the corresponding lab parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 12 | 15 | 2
Participants
  Anemia: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 10 | 15 | 2
  Anemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  INR increased: number analyzed (Participants) | 2 | 2 | 2 | 4 | 14 | 15 | 6 | 5 | 12 | 10 | 13 | 2
  INR increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocyte count decreased: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 4 | 13 | 10 | 15 | 2
  Lymphocyte count decreased | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 2 | 2 | 0 | 0
  Neutrophil count decreased: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 13 | 10 | 15 | 2
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
  White blood cell decreased: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 10 | 15 | 2
  White blood cell decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Laboratory Abnormalities-Chemistries
Description: Participants who experienced chemistry laboratory test abnormalities were summarized according to worst toxicity grade observed for each chemistry laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03 (Grade 0: no change from normal or reference range; Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated). This outcome measure calculated the number of participants with chemistry laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above, including the following parameters: alanine aminotransferase (ALT) increased, alkaline phosphatase (ALP) increased, aspartate aminotransferase (AST) increased, hyperglycemia, hypermagnesemia, hypocalcemia, hypokalemia, hyponatremia, hypophosphatemia, lipase increased, serum amylase increased.
Time Frame: as for outcome 4
Population: Participants who had at least one on-treatment assessment for the corresponding lab parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 12 | 15 | 2
Participants
  ALT increased: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 10 | 15 | 2
  ALT increased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  ALP increased: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 10 | 15 | 2
  ALP increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AST increased: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 10 | 15 | 2
  AST increased | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Hyperglycemia: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 10 | 15 | 2
  Hyperglycemia | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Hypermagnesemia: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 13 | 10 | 15 | 2
  Hypermagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypocalcemia: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 12 | 9 | 15 | 2
  Hypocalcemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypokalemia: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 10 | 15 | 2
  Hypokalemia | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Hyponatremia: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 10 | 15 | 2
  Hyponatremia | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 3 | 1 | 0 | 0
  Hypophosphatemia: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 13 | 10 | 15 | 2
  Hypophosphatemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
  Lipase increased: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 12 | 10 | 15 | 2
  Lipase increased | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0
  Serum amylase increased: number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 13 | 10 | 15 | 2
  Serum amylase increased | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Laboratory Abnormalities-Urinalysis
Description: Participants who experienced urinalysis laboratory test abnormalities were summarized according to worst toxicity grade observed for each urinalysis laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03 (Grade 0: no change from normal or reference range; Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated). This outcome measure calculated the number of participants with urinalysis laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above.
Time Frame: as for outcome 4
Population: Participants who had at least one on-treatment assessment for the corresponding lab parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 14 | 15 | 6 | 4 | 3 | 6 | 6 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Vital Signs Data Meeting Pre-Defined Criteria
Description: Blood pressure (BP), including systolic BP (SBP) and diastolic BP (DBP), and pulse rate were recorded in a supine or seated position.
Time Frame: From baseline up to follow up (at least 28 days and no more than 35 days after discontinuation of treatment), maximum treatment duration: 89.3 weeks for Part 1A, 49.4 weeks for Part 2A, 53.7 weeks for Part 1B
Population: Participants who were evaluated against criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 5 | 14 | 12 | 15 | 2
Participants
  Pulse rate >120 beats per minute (bpm) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 3 | 2 | 1 | 0
  Increase in SBP ≥30 mmHg | 0 | 0 | 2 | 2 | 2 | 9 | 1 | 1 | 3 | 3 | 4 | 1
  Decrease in SBP ≥30 mmHg | 0 | 1 | 0 | 2 | 4 | 5 | 0 | 3 | 1 | 1 | 1 | 0
  Increase in DBP ≥20 mmHg | 0 | 0 | 2 | 2 | 3 | 7 | 2 | 2 | 2 | 4 | 5 | 1
  Decrease in DBP ≥20 mmHg | 0 | 1 | 0 | 1 | 4 | 6 | 0 | 2 | 1 | 1 | 0 | 0
  SBP value <90 mmHg | 0 | 0 | 0 | 0 | 2 | 6 | 0 | 1 | 2 | 0 | 0 | 0
  DBP value <50 mmHg | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 1 | 0 | 0

8. Primary Outcome: Percentage of Participants With Objective Response in Part 2
Description: Percentage of participants with objective response based on assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 6 weeks from the start of treatment until disease progression, death, or permanent discontinuation of study treatment (maximum treatment duration: 49.4 weeks)
Population: Participants received at least 1 dose of study treatment with adequate baseline assessment and at least 1 determinate post baseline assessment, disease progression, or death before the first tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC
Number analyzed (Participants) | 4 | 11 | 10 | 11
Percentage of participants | 25.0 [0.6 to 80.6] | 45.5 [16.7 to 76.6] | 10.0 [0.3 to 44.5] | 27.3 [6.0 to 61.0]

9. Primary Outcome: Duration of Response (DR) in Part 2
Description: Duration of response (DR) was the time from first documentation of PR or CR to date of first documentation of progressive disease (PD) or death due to any cause. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of one or more new lesions.
Time Frame: as for outcome 8
Population: Participants received at least 1 dose of study treatment with adequate baseline assessment and at least 1 determinate post baseline assessment, disease progression, or death before the first tumor assessment. DR was only for the subset participants with an objective response.
Measure: Median (95% Confidence Interval); unit: Month
Groups:
- PART 2A PF-06804103 3.0 mg/kg HER2+ BC: Participants with HER2-positive BC in 3L setting received PF-06804103 at 3.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 2A was approximately 49.4 weeks.
- PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC: Participants with HR-positive HER2 IHC
  1+ or IHC 2+/ISH- BC in 2L setting received PF-06804103 at 3.0 mg/kg on Day 1 of each 21-day cycle as an IV infusion. The maximum duration of treatment for Part 2A was approximately 49.4 weeks.
Arm/Group | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC
Number analyzed (Participants) | 1 | 5 | 1 | 3
Month | NA [NA to NA] — Because there were few confirmed responders for specific treatment groups and the duration of response was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | 2.9 [2.4 to NA] — Because there were few confirmed responders for specific treatment groups and the duration of response was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | 4 [NA to NA] — Because there were few confirmed responders for specific treatment groups and the duration of response was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | NA [4.4 to NA] — Because there were few confirmed responders for specific treatment groups and the duration of response was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible.

10. Primary Outcome: Progression-Free Survival (PFS) in Part 2
Description: Progression-free survival (PFS) was the time from randomization date to date of first documentation of PD or death due to any cause. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of one or more new lesions.
Time Frame: as for outcome 8
Population: All enrolled participants in part 2A.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC
Number analyzed (Participants) | 5 | 14 | 12 | 15
Month | NA [2.6 to NA] — Because the number of participants in specific treatment groups is small and the PFS was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | 5.5 [2.9 to NA] — Because the number of participants in specific treatment groups is small and the PFS was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | 1.3 [0.7 to 6.4] | 5.6 [2.4 to NA] — Because the number of participants in specific treatment groups is small and the PFS was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible.

11. Primary Outcome: Time to Tumor Progression (TTP) in Part 2
Description: Time to progression (TTP) was the time from start date to the date of the first documentation of PD. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of one or more new lesions.
Time Frame: Baseline, every 6 weeks from the start of treatment until disease progression, death, or withdrawal from treatment (maximum treatment duration: 49.4 weeks)
Population: All enrolled participants in part 2A.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC
Number analyzed (Participants) | 5 | 14 | 12 | 15
Month | NA [2.6 to NA] — Because the number of participants in specific treatment groups is small and the TTP was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | 5.5 [2.9 to NA] — Because the number of participants in specific treatment groups is small and the TTP was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | 1.3 [0.7 to NA] — Because the number of participants in specific treatment groups is small and the TTP was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | 5.6 [2.4 to NA] — Because the number of participants in specific treatment groups is small and the TTP was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible.

12. Secondary Outcome: Percentage of Participants With Objective Response in Part 1
Description: as for outcome 8
Time Frame: Baseline, every 6 weeks (for Part 1A) or every 8 weeks (for Part 1B) from the start of treatment until disease progression, death, or permanent discontinuation of study treatment (maximum treatment duration: 89.3 weeks for Part 1A, 53.7 weeks for Part 1B)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PART 1A PF- 06804103 < 2.0 mg/kg: Participants with HER2-positive BC or HER-positive GC received PF-06804103 at 0.15 mg/kg or 0.5 mg/kg or 1.2 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06804103 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment for part 1A was approximately 89.3 weeks.
Arm/Group | PART 1A PF- 06804103 < 2.0 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 6 | 4 | 14 | 14 | 5 | 1
Percentage of participants | 16.7 [0.4 to 64.1] | 0 [0.0 to 60.2] | 21.4 [4.7 to 50.8] | 42.9 [17.7 to 71.1] | 60.0 [14.7 to 94.7] | 100.0 [2.5 to 100.0]

13. Secondary Outcome: Duration of Response (DR) in Part 1
Description: as for outcome 9
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Month
Groups:
- PART 1A PF-06804103 0.15 mg/kg: Participants with HER2-positive BC or HER2-positive GC received PF-06804103 at 0.15 mg/kg on Day 1 of each 21-day cycle as an intravenous (IV) infusion. The maximum duration of treatment for Part 1A was approximately 89.3 weeks.
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 3 | 6 | 3 | 1
Month |  |  | 4.2 [NA to NA] — Because there were no or few confirmed responders for specific treatment groups and the duration of response was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. |  | 15.5 [6 to 18.9] | 7.3 [5.5 to 18.7] | NA [NA to NA] — Because there were no or few confirmed responders for specific treatment groups and the duration of response was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | NA [NA to NA] — Because there were no or few confirmed responders for specific treatment groups and the duration of response was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible.

14. Secondary Outcome: Progression-Free Survival (PFS) in Part 1
Description: as for outcome 10
Time Frame: as for outcome 12
Population: All enrolled participants in part 1.
Measure: Median (95% Confidence Interval); unit: Month
Groups:
- PART 1A PF-06804103 < 2.0 mg/kg: Participants with HER2-positive BC or HER-positive GC received PF-06804103 at 0.15 mg/kg or 0.5 mg/kg or 1.2 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06804103 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment for part 1A was approximately 89.3 weeks.
Arm/Group | PART 1A PF-06804103 < 2.0 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 6 | 4 | 16 | 15 | 6 | 2
Month | 4.2 [0.7 to 15.7] | 3.4 [2.6 to NA] — Because the number of participants in specific treatment groups is small and the PFS was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | 4.7 [1.2 to 7.2] | 8.2 [4.3 to 14.9] | NA [2.7 to NA] — Because the number of participants in specific treatment groups is small and the PFS was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | NA [NA to NA] — Because the number of participants in specific treatment groups is small and the PFS was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible.

15. Secondary Outcome: Time to Tumor Progression (TTP) in Part 1
Description: as for outcome 11
Time Frame: as for outcome 12
Population: All enrolled participants in part 1.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | PART 1A PF-06804103 < 2.0 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 6 | 4 | 16 | 15 | 6 | 2
Month | 4.2 [0.7 to 15.7] | 3.4 [2.6 to NA] — Because the number of participants in specific treatment groups is small and the TTP was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | 4.7 [1.2 to 7.2] | 8.2 [4.3 to 14.9] | NA [2.7 to NA] — Because the number of participants in specific treatment groups is small and the TTP was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible. | NA [NA to NA] — Because the number of participants in specific treatment groups is small and the TTP was censored for some participants, therefore there were insufficient number of participants with events, the estimation of median and 95% confidence intervals may not be feasible.

16. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibody (NAb) Against PF-06804103
Description: To evaluate the immunogenicity as measured by presence of ADA and NAb in participants treated with PF-06804103.
Time Frame: Prior to the start of treatment on Day 1 of Cycle 1 up to end of treatment (maximum treatment duration: 89.3 weeks for Part 1A, 49.4 weeks for Part 2A, 53.7 weeks for Part 1B)
Population: All enrolled participants who received at least one dose of study treatment and had at least 1 ADA sample collected.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 12 | 15 | 6 | 5 | 13 | 10 | 15 | 2
Participants
  Participants with ADA | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 2 | 4 | 5 | 0
  Participants with NAb | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0

17. Secondary Outcome: Number of Participants With HER2 Positivity Based on Tumor Tissue Analysis
Description: Tumor tissues from archived tissue biopsy were analyzed for HER2 mutations.
Time Frame: Baseline
Population: All enrolled participants with at least 1 of the biomarkers evaluated at pre- and/or post-dose.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 14 | 15 | 6 | 5 | 14 | 12 | 15 | 2
Participants | 2 | 2 | 1 | 3 | 10 | 13 | 6 | 5 | 14 | 4 | 1 | 0

18. Secondary Outcome: Maximum Observed Concentration (Cmax) of PF-06804103 Antibody-Drug Conjugate (ADC)
Description: Cmax is maximum observed serum concentration. Cmax for PF-06804103 ADC was observed directly from data. Part 2A used a sparse pharmacokinetic (PK) sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: Pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose of Cycle 1 & 4 Day 1 for Part 1A; pre-dose, 1, 4, 24, 72, 168 hours post-dose of Cycle 1 & 4 Day 1 for Part 1B
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
microgram/milliliter (µg/mL)
  Cycle 1 | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 36.97 (24) | 71.24 (21) | 78.91 (21) | 103.1 (28) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
  Cycle 4 |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 43.00 (15) | 53.29 (29) | 76.52 (24) | 82.13 (7) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

19. Secondary Outcome: Terminal Serum Half-Life (t1/2) of PF-06804103 ADC
Description: Terminal serum half-life (t1/2) is the time measured for the serum concentration of drug to decrease by one half. Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: as for outcome 18
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
Day
  Cycle 1 | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.495 (0.76081) | 4.257 (1.1289) | 5.001 (1.2963) | 4.962 (1.3623) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
  Cycle 4 |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4.177 (1.1648) | 5.185 (1.1855) | 5.278 (2.2199) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

20. Secondary Outcome: Area Under The Serum Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06804103 ADC
Description: AUCinf is the area under the serum concentration-time profile from time zero extrapolated to infinite time. Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: Pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose of Cycle 1 Day 1 for Part 1A; pre-dose, 1, 4, 24, 72, 168 hours post-dose of Cycle 1 Day 1 for Part 1B
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (µg*hr/mL)
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
microgram*hour/milliliter (µg*hr/mL) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 5120 (11) | 9498 (32) | 12940 (31) | 16550 (38) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

21. Secondary Outcome: Area Under the Concentration-Time Profile From Time Zero to Time Tau (AUCtau) of PF-06804103 ADC
Description: Tau refers to the dosing interval and it equals to 504 hours for Part 1A and 336 hours for Part 1B. AUCtau is the area under the concentration-time profile from time zero to time tau. AUCtau for PF-06804103 ADC was determined using linear/log trapezoidal method. Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: Pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose of Cycle 4 Day 1 for Part 1A; pre-dose, 1, 4, 24, 72, 168 hours post-dose of Cycle 4 Day 1 for Part 1B
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
µg*hr/mL |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 7504 (28) | 10730 (33) | 11990 (23) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

22. Secondary Outcome: Clearance (CL) of PF-06804103 ADC
Description: Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance for PF-06804103 ADC was calculated as dose/AUCinf for single dose and dose/AUCtau for multiple dose, where AUCinf was the area under the serum concentration-time profile from time zero extrapolated to infinite time and AUCtau was the area under the concentration-time profile from time zero to time tau (tau equals to 504 hours for Part 1A and 336 hours for Part 1B). Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: as for outcome 18
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/hr)
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
Liter/hour (L/hr)
  Cycle 1 | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.02073 (32) | 0.01970 (27) | 0.01884 (24) | 0.01975 (40) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
  Cycle 4 |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.02069 (28) | 0.01731 (27) | 0.01971 (49) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

23. Secondary Outcome: Volume of Distribution at Steady State (Vss) of PF-06804103 ADC
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state. Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: as for outcome 21
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
Liter (L) |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.037 (15) | 3.106 (24) | 3.467 (24) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

24. Secondary Outcome: Observed Accumulation Ratio (Rac) of PF-06804103 ADC
Description: Rac is defined as observed accumulation ratio based on dose normalized AUCtau (AUCtau[dn]), where AUCtau is the area under the concentration-time profile from time zero to time tau (tau equals to 504 hours for Part 1A and 336 hours for Part 1B). Rac=[Cycle 4 Day 1 AUCtau(dn) (multiple dose)] /[Cycle 1 Day 1 AUCtau(dn) (single Dose)] for Part 1A, Rac=[Cycle 3 Day 1 AUCtau(dn) (multiple dose)] /[Cycle 1 Day 1 AUCtau(dn) (single Dose)] for Part 1B. Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: Pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose of Cycle 1 & 4 Day 1 for Part 1A; pre-dose, 1, 4, 24, 72, 168 hours post-dose of Cycle 1 Day 1, pre-dose, 1 hour post-dose of Cycle 3 Day 1 for Part 1B
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
Ratio |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1.007 (20) | 1.164 (22) | 1.114 (15) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

25. Secondary Outcome: Cmax of PF-06804103 Total Antibody
Description: Cmax is maximum observed serum concentration. Cmax for PF-06804103 total antibody was observed directly from data. Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure. Total antibody means PF-06804103 with or without PF-06380101 conjugated. Both the antibody and small molecule components of the ADC are critical to its activity, requiring assays suited to measuring these disparate components. Each analyte provides unique information regarding ADC behavior in vivo and, singly or in combination, facilitates understanding of ADC PK.
Time Frame: as for outcome 18
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
µg/mL
  Cycle 1 | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 46.77 (24) | 78.17 (34) | 89.67 (31) | 117.7 (19) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
  Cycle 4 |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 44.02 (10) | 59.96 (26) | 77.53 (21) | 88.54 (9) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

26. Secondary Outcome: t1/2 of PF-06804103 Total Antibody
Description: as for outcome 19
Time Frame: as for outcome 18
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
Day
  Cycle 1 | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4.438 (2.3541) | 4.775 (2.3152) | 5.679 (2.4450) | 4.530 (1.1946) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
  Cycle 4 |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.520 (0.45133) | 4.188 (1.1884) | 5.159 (1.0528) | 5.423 (3.3577) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

27. Secondary Outcome: AUCinf of PF-06804103 Total Antibody
Description: as for outcome 20
Time Frame: as for outcome 20
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
µg*hr/mL | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 6868 (62) | 10770 (53) | 15360 (58) | 18010 (38) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

28. Secondary Outcome: AUCtau of PF-06804103 Total Antibody
Description: Tau refers to the dosing interval and it equals to 504 hours for Part 1A and 336 hours for Part 1B. AUCtau is the area under the concentration-time profile from time zero to time tau. AUCtau for PF-06804103 total antibody was determined using linear/log trapezoidal method. Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: as for outcome 21
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
µg*hr/mL |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4826 (18) | 8231 (30) | 10980 (32) | 12870 (21) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

29. Secondary Outcome: CL of PF-06804103 Total Antibody
Description: Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance for PF-06804103 total antibody was calculated as dose/AUCinf for single dose and dose/AUCtau for multiple dose, where AUCinf was the area under the serum concentration-time profile from time zero extrapolated to infinite time and AUCtau was the area under the concentration-time profile from time zero to time tau (tau equals to 504 hours for Part 1A and 336 hours for Part 1B). Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: as for outcome 18
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
L/hr
  Cycle 1 | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.01544 (103) | 0.01737 (47) | 0.01587 (46) | 0.01899 (37) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
  Cycle 4 |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.01777 (15) | 0.01890 (29) | 0.01693 (27) | 0.02023 (37) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

30. Secondary Outcome: Vss of PF-06804103 Total Antibody
Description: as for outcome 23
Time Frame: as for outcome 21
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
L |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.180 (9) | 2.781 (12) | 3.011 (23) | 3.520 (20) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

31. Secondary Outcome: Rac of PF-06804103 Total Antibody
Description: as for outcome 24
Time Frame: as for outcome 24
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
Ratio |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.7427 (73) | 1.033 (18) | 1.097 (15) | 1.122 (19) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

32. Secondary Outcome: Cmax of PF-06380101 Unconjugated Payload
Description: Cmax is maximum observed serum concentration. Cmax for PF-06380101 unconjugated payload was observed directly from data. Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure. Small molecule components (PF-06380101) of the ADC are critical to its activity, requiring assays suited to measuring these disparate components. Each analyte provides unique information regarding ADC behavior in vivo and, singly or in combination, facilitates understanding of ADC PK.
Time Frame: as for outcome 18
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
nanogram/milliliter (ng/mL)
  Cycle 1 | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1.706 (73) | 3.180 (41) | 4.219 (43) | 6.916 (67) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
  Cycle 4 |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.254 (108) | 2.185 (59) | 3.094 (78) | 4.790 (15) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

33. Secondary Outcome: Time for Cmax (Tmax) of PF-06380101 Unconjugated Payload
Description: Tmax is the time for Cmax. Tmax for PF-06380101 unconjugated payload was observed directly from data as time of first occurrence.Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: as for outcome 18
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: Hour
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
Hour
  Cycle 1 | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 117 [69.0 to 187] | 71.7 [22.6 to 169] | 143 [48.0 to 192] | 93.5 [68.0 to 192] | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
  Cycle 4 |  | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 70.1 [43.9 to 73.3] | 140 [47.9 to 167] | 105 [46.1 to 166] | 84.0 [69.0 to 96.0] | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

34. Secondary Outcome: t1/2 of PF-06380101 Unconjugated Payload
Description: as for outcome 19
Time Frame: as for outcome 18
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
Day
  Cycle 1 | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4.170 (0.55923) | 4.384 (1.1479) | 5.164 (1.2816) | 4.795 (1.3663) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
  Cycle 4 |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4.723 (0.35275) | 5.214 (1.0385) | 5.889 (1.4216) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

35. Secondary Outcome: AUCinf of PF-06380101 Unconjugated Payload
Description: as for outcome 20
Time Frame: as for outcome 20
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 16 | 15 | 6 | 2
nanogram*hour/milliliter (ng*hr/mL) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 465.8 (45) | 945.4 (51) | 1256 (43) | 1824 (83) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

36. Secondary Outcome: AUCtau of PF-06380101 Unconjugated Payload
Description: as for outcome 28
Time Frame: as for outcome 21
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
ng*hr/mL |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 478.0 (124) | 556.5 (45) | 780.8 (56) | 1136 (19) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

37. Secondary Outcome: Rac of PF-06380101 Unconjugated Payload
Description: Rac is defined as observed accumulation ratio based on dose normalized AUCtau (AUCtau[dn]), where AUCtau is the area under the concentration-time profile from time zero to time tau (tau equals to 504 hours for Part 1A and 336 hours for Part 1B). Rac=[Cycle 4 Day 1 AUCtau(dn) (multiple dose)]/[Cycle 1 Day 1 AUCtau(dn) (single Dose)] for Part 1A, Rac=[Cycle 3 Day 1 AUCtau(dn) (multiple dose)]/[Cycle 1 Day 1 AUCtau(dn) (single Dose)] for Part 1B. Part 2A used a sparse PK sampling schedule leaving very limited data for PK parameter estimation, so PK parameters from Part 2A were not reported. Only part 1A and part 1B treatment groups were included in this outcome measure.
Time Frame: as for outcome 24
Population: Participants who received at least 1 dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 9 | 12 | 4 | 1
Ratio |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1.083 (64) | 0.8088 (28) | 0.9427 (49) | 0.8507 (35) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last treatment administration, maximum duration between first and last dose: 89.3 weeks for Part 1A, 49.4 weeks for Part 2A, 53.7 weeks for Part 1B
Description: MedDRA 24.1 coding dictionary was applied for all AE tables. The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PART 1A PF-06804103 0.15 mg/kg | PART 1A PF-06804103 0.5 mg/kg | PART 1A PF-06804103 1.2 mg/kg | PART 1A PF-06804103 2.0 mg/kg | PART 1A PF-06804103 3.0 mg/kg | PART 1A PF-06804103 4.0 mg/kg | PART 1A PF-06804103 5.0 mg/kg | PART 2A PF-06804103 3.0 mg/kg HER2+ BC | PART 2A PF-06804103 4.0 mg/kg HER2+ BC | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/2 | 0/2 | 1/4 | 0/16 | 1/15 | 1/6 | 0/5 | 0/14 | 3/12 | 1/15 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2 | 0/2 | 1/4 | 7/16 | 5/15 | 4/6 | 2/5 | 6/14 | 5/12 | 7/15 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 4/4 | 16/16 | 15/15 | 6/6 | 5/5 | 14/14 | 11/12 | 15/15 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PART 1A PF-06804103 0.15 mg/kg (N=2) | PART 1A PF-06804103 0.5 mg/kg (N=2) | PART 1A PF-06804103 1.2 mg/kg (N=2) | PART 1A PF-06804103 2.0 mg/kg (N=4) | PART 1A PF-06804103 3.0 mg/kg (N=16) | PART 1A PF-06804103 4.0 mg/kg (N=15) | PART 1A PF-06804103 5.0 mg/kg (N=6) | PART 2A PF-06804103 3.0 mg/kg HER2+ BC (N=5) | PART 2A PF-06804103 4.0 mg/kg HER2+ BC (N=14) | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC (N=12) | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC (N=15) | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC (N=2)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PART 1A PF-06804103 0.15 mg/kg (N=2) | PART 1A PF-06804103 0.5 mg/kg (N=2) | PART 1A PF-06804103 1.2 mg/kg (N=2) | PART 1A PF-06804103 2.0 mg/kg (N=4) | PART 1A PF-06804103 3.0 mg/kg (N=16) | PART 1A PF-06804103 4.0 mg/kg (N=15) | PART 1A PF-06804103 5.0 mg/kg (N=6) | PART 2A PF-06804103 3.0 mg/kg HER2+ BC (N=5) | PART 2A PF-06804103 4.0 mg/kg HER2+ BC (N=14) | PART 2A PF-06804103 3.0 mg/kg HR+ HER2-Low BC (N=12) | PART 2A PF-06804103 4.0 mg/kg HR+ HER2-Low BC (N=15) | PART 1B PF-06804103 2.0 mg/kg HR+ HER2-Low Combo BC (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 7 | 3 | 2 | 0 | 4 | 3 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corneal disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 2 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid rash (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Keratopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Visual brightness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 6 | 1 | 0 | 1 | 3 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 5 | 4 | 4 | 2 | 3 | 5 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 4 | 2 | 1 | 1 | 0 | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4 | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 4 | 4 | 2 | 0 | 4 | 3 | 4 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 4 | 2 | 1 | 4 | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 5 | 1 | 0 | 0 | 1 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 2 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 2 | 10 | 6 | 5 | 2 | 5 | 5 | 2 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 4 | 2 | 0 | 1 | 2 | 1 | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blister infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 2 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Cystitis escherichia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pustule (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 3 | 4 | 1 | 1 | 3 | 2 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Human epidermal growth factor receptor decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 0
Lung diffusion test decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Total lung capacity abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 2 | 3 | 8 | 3 | 1 | 5 | 2 | 3 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 4 | 6 | 2 | 2 | 2 | 3 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 3 | 3 | 3 | 0 | 2 | 0 | 5 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 3 | 2 | 3 | 0 | 2 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 4 | 1 | 1 | 3 | 6 | 7 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 5 | 5 | 2 | 0 | 6 | 4 | 5 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 8 | 3 | 3 | 0 | 1 | 2 | 4 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 1 | 1 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 3 | 6 | 2 | 1 | 7 | 4 | 5 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vocal cord paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 1 | 2 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 3 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 4 | 10 | 3 | 1 | 5 | 6 | 9 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 2 | 2 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nodular rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 3 | 1 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 5 | 2 | 2 | 7 | 4 | 3 | 2
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 3 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
On 10 February 2021, a decision was made by the sponsor to terminate the study due to business reasons. The decision was not due to any urgent patient safety concerns, study conduct issues, or regulatory authority requests concerning treatment with the PF-06804103 compound. Part 2B had not enrolled prior to the termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT03284723/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03284723/SAP_001.pdf